CLINICAL TRIAL: NCT00550407
Title: Study SCA104779, an Evaluation of BW430C (Lamotrigine) Versus Placebo in the Prevention of Mood Episodes in Bipolar I Disorder Patients
Brief Title: An Evaluation Of BW430C (Lamotrigine) Versus Placebo In The Prevention Of Mood Episodes In Bipolar I Disorder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCA104779
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Results first posted 2010-07-27 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Bipolar Disorder
Keywords: Lamotrigine; Prevention of relapse or recurrence of a mood episode; Bipolar I disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BW430C(lamotrigine) (Active Comparator)
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — lamotrigine 100mg/day or 200mg/day
  Arms: BW430C(lamotrigine)
Drug: Placebo — placebo once daily
  Arms: Placebo

SUMMARY:
This study is planned to objectively assess the efficacy and safety of lamotrigine maintenance therapy after symptoms of mood episode had been stabilised by open-label treatment with lamotrigine alone or in combination with other psychotropic medication in patients with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

At Screening Disease to be studied: Has a diagnosis of following disease as defined by DSM-IV-TR criteria.

* Bipolar I Disorder, most recent episode depressed（296.5x）
* Bipolar I Disorder, most recent episode hypomanic（296.40）
* Bipolar I Disorder, most recent episode manic（296.4x） The diagnosis of mood episode will be made with reference to Mini International Neuropsychiatric Interview: M.I.N.I, Japanese Version.

At Screening

The subject who has a diagnose of bipolar I disorder, most recent episode depressed (296.5x) must meet the following criteria:

* Is currently experiencing a major depressive episode or has had a major depressive episode as defined by DSM-IV-TR criteria within 60 days of the screening visit and at least one additional major depressive episode and one manic or hypomanic episode, as defined by DSM-IV-TR criteria, within 3 years of enrolment. A well documented history of a mixed episode that meets DSM-IV-TR criteria may be counted as a previous episode.All subjects must have experienced at least one well-documented manic or mixed episode in the past.
* Has a duration of the most recent/current depressive episode of at least 2 weeks but not longer than 12 months prior to enrolment.
* The subject without current major depressive episode must have a major depressive episode within 60 days of screening and has depressive symptoms at screening or is under treatment for depressive symptoms, which can be confirmed by medical record, etc.
* If the subject is currently experiencing a major depressive episode, the subject must have a minimum total score on the HAM-D (17-item scale) of 18 at the screening. This criterion will not apply to the subject with recent depressive episode.

At Screening

The subject who has a diagnose of bipolar I disorder, most recent episode hypomanic（296.4x） or bipolar I disorder, most recent episode manic（296.5x） must meet the following criteria:

* Has experienced a recent manic or hypomanic episode (current or within 60 days of the Screening Visit) and has had at least one additional manic or hypomanic episode and one depressed episode, as defined by DSM-IV-TR criteria, within three years of enrolment. A well documented history of a mixed episode that meets DSM-IV-TR criteria may be counted as a previous episode. All subjects must have experienced at least one well-documented manic or mixed episode in the past.
* Has a duration of the index manic episode of at least 1 week (unless hospitalised) or hypomanic episode of at least 4 days. In neither case should the index episode be more than 12 months in duration.
* The subject current experiencing hypomania episode or without current episode must have a manic episode which can be confirmed by medical record, etc. The subject without current episode must have a episode within 60 days of screening and has manic or hypomanic symptomatology is under treatment for manic or hypomanic symptoms.
* If the subject's index episode is subject initial manic mood event, subject must have a minimum score of 10 (moderate severity) on the first 11 items of the YMRS at the screening. A threshold YMRS score that indicates significant manic symptoms is not required for patients who previously experienced well-documented DSM-IV-level mania or when the index episode is hypomania or when a subject's index manic or hypomanic episode is documented to have occurred within 60 days of the screening Visit.

At Screening Age: Is at least 20 years of age (at the time of informed consent). At Screening Sex: either sex. Female of child-bearing potential will be eligible for inclusion in this study. However they have to have a negative pregnancy test at the screening visit, agree to further pregnancy testing at the time points determined in study assessments and procedures and practice one of the following methods of contraception from the screening visit until the end of the follow-up examination.

* Abstinence
* Injectable progestogen
* Implants of levonorgestrel
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Double barrier method: condom or occlusive cap (diaphragm or cervical / vault caps) plus spermicidal agent (foam /gel / film / cream / suppository) At Screening In/Out patient: Either At Screening Informed consent: the subject capable of giving written informed consent. At Week 0 of First Phase (titration) If the subject is currently experiencing a major depressive episode, the subject must have a minimum total score at baseline on the HAM-D (17-item scale) of 18 at the start of First Phase. This criterion will not apply to the subject with recent depressive episode.

At Week 0 of First Phase (titration) If the subject's index episode is subject initial manic mood event, subject must have a minimum total score at baseline of 10 (moderate severity) on the first 11 items of the YMRS at the start of First Phase (titration). A threshold YMRS score that indicates significant manic symptoms is not required for patients who previously experienced well-documented DSM-IV-level mania or when the index episode is hypomania or when a subject's index manic or hypomanic episode is documented to have occurred within 60 days of the screening Visit.

At Week 0 of Second Phase (maintenance therapy) Each subject completing 8 to 16 weeks of open-label lamotrigine treatment in the First Phase must meet all of the following inclusion criteria to be eligible for entry into the Second Phase (maintenance therapy, randomization phase).

At Week 0 of Second Phase (maintenance therapy) Has no tolerability problem with lamotrigine at a minimum dosage of 100 mg/day during the final 2 weeks of the First Phase (titration).

At Week 0 of Second Phase (maintenance therapy) Has improved/stabilised during the First Phase (titration) as indicated by a CGI-S score of ≤3 (mildly ill). Once improved, the subject must also demonstrate sustained improvement by achieving a CGI-S score of ≤3 (mildly ill) for at least 4 consecutive weeks of treatment immediately prior to the Second Phase (maintenance therapy) (randomization).

At Week 0 of Second Phase (maintenance therapy) Has demonstrated adequate compliance with the study treatment in the First Phase (titration) (compliance rate: at least 70%).

At Week 0 of Second Phase (maintenance therapy) In/Out patient: Either

Exclusion Criteria:

At Screening Has a DSM-IV-TR diagnosis of rapid cycling and has had more than six mood episodes including depression, mania, hypomania or mixed, in the 12-month period prior to screening. Note: while 4 or more episodes in the past 12 months constitute rapid cycling up to six episodes in the past 12 months are allowed in this protocol.

At Screening Has a DSM-IV-TR diagnosis of bipolar I disorder, most recent episode mixed (296.6x).

At Screening Has a DSM-IV-TR diagnosis of Axis II which would suggest non-responsiveness to pharmacotherapy for bipolar disorder.

At Screening Has a DSM-IV-TR diagnosis of or has received treatment for major depressive disorder, panic disorder, obsessive-compulsive disorder, social phobia, bulimia nervosa, schizophrenia or schizoaffective disorder within 12 months of screening.

At Screening Has a history of substance (including alcohol and drugs) dependence within 12 months of screening or abuse within 1 month of screening according to DSM-IV-TR.

At Screening Patients whose mood episode is due to direct physiological effects of a general medical condition (for example, hypothyroidism, hyperthyroidism) At Screening Has a score of 3 or more on item of the HAM-D related to suicide or is at a high suicidal risk in the judgment of the investigator/sub-investigator.

At Screening Has a history of severe rash or rash due to anti-epileptic drugs. At Screening Patients with severe hepatic/renal/cardiac/pulmonary disorder or hematopoietic disorder. The severity refers to Grade 3 according to the Classification of the Severity of Adverse Experiences (PAB/SD Notification No. 80, dated 29 June 1992).

At Screening Patients have less than 5 years of remission history from clinically significant malignancy (other than e.g. basal cell or squamous cell skin cancer, in-situ carcinoma of cervix or prostate CA in situ).

At Screening Patients with chronic hepatitis typeB and /or typeC which is positive of hepatitis B surface antigen （HBsAg）and/or hepatitis C antibody.

At Screening Has an acute or chronic illness likely to impair drug absorption, distribution, metabolism or excretion or has any unstable physical symptoms likely to require hospitalisation during participation in the study.

At Screening Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study.

At Screening Has a history or current diagnosis of epilepsy. At Screening Has a history of treatment with lamotrigine. At Screening Patients with a history of drug allergy to any ingredient of the test-drug. At Screening Has received an investigational drug within 30 days of screening. At Screening Is morbidly obese (Body Mass Index [BMI] >40) BMI = body weight (kg)/height (m2).

At Screening Patients whom the investigator or sub-investigator considers ineligible for the study.

At Week 0 of First Phase (titration) Has a score of 3 or more on item of the HAM-D related to suicide or is at a high suicidal risk in the judgment of the investigator/sub-investigator and continues .to meet the criteria at the screening visit.

At Week 0 of Second Phase (maintenance therapy) Has signs or symptoms of psychosis. At Week 0 of Second Phase (maintenance therapy) Has a score of 3 or more on item of the HAM-D related to suicide or is at a high suicidal risk in the judgment of the investigator/sub-investigator.

At Week 0 of Second Phase (maintenance therapy) Has had a change in lamotrigine dosage during the final week of the First Phase (titration).

At Week 0 of Second Phase (maintenance therapy) Has a diagnosis of bipolar I disorder, most recent episode of depressed (296.5x) and has experienced manic, hypomanic or mixed symptoms; Has a diagnosis of bipolar I disorder, most recent episode hypomanic (296.40) or most recent episode manic (296.4x) and has experienced depressive symptoms, that require treatment during the First Phase (titration).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Japan (20):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tsukasa Koyama, Teruhiko Higuchi, Shigeto Yamawaki, Shigenobu Kanba, Takeshi Terao, Atsuko Shinohara. Study SCA104779, an evaluation of BW430C (lamotrigine) versus placebo in the prevention of mood episodes in bipolar I disorder patients. Japanese Journal of Clinical Psychiatry. 2011;40(3):369-383.
- [Derived] Hashimoto Y, Kotake K, Watanabe N, Fujiwara T, Sakamoto S. Lamotrigine in the maintenance treatment of bipolar disorder. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD013575. doi: 10.1002/14651858.CD013575.pub2. PMID 34523118
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: SCA104779 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCA104779 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA104779 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA104779 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants whose symptoms of mood episodes were stabilized with lamotrigine in the Preliminary Phase (Clinical Global Impressions of Severity score of 3 [mild] or less for at least 4 consecutive weeks, and lamotrigine given as monotherapy for at least 1 week before the start of the Randomized Phase) were randomized to placebo or lamotrigine.
Groups:
- Lamotrigine 25-200 mg: The dose of lamotrigine was increased gradually in the dose range of 25-200 milligrams (mg)/day, while the doses of other medications for bipolar disorder were decreased gradually
- Placebo: Matching placebo
- Lamotrigine 200 mg: Lamotrigine 200 mg once a day. The dose may have been reduced to 100 mg/day for safety reasons at the discretion of the investigator/subinvestigator. The use of other medications for bipolar disorder was prohibited.
Period: 8-16 Week Preliminary (Open-Label) Phase
Arm/Group | Lamotrigine 25-200 mg | Placebo | Lamotrigine 200 mg
Started | 215 | 0 | 0
Completed | 103 | 0 | 0
Not Completed | 112 | 0 | 0
Not completed — Adverse Event | 55 | 0 | 0
Not completed — Lack of Efficacy | 39 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Defined Stopping Criteria Reached | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Investigator Discretion | 8 | 0 | 0
Not completed — Withdrew Consent | 6 | 0 | 0
Not completed — Continuation Criteria Not Met | 1 | 0 | 0
Period: 26-Week Randomized Phase
Arm/Group | Lamotrigine 25-200 mg | Placebo | Lamotrigine 200 mg
Started | 0 | 58 | 45
Completed | 0 | 15 | 21
Not Completed | 0 | 43 | 24
Not completed — Adverse Event | 0 | 5 | 2
Not completed — Lack of Efficacy | 0 | 36 | 19
Not completed — Investigator Discretion | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lamotrigine 200 mg | Total
Number analyzed (Participants) | 58 | 45 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (12.68) | 42.4 (11.79) | 42.8 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 27 | 18 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese Heritage | 58 | 44 | 102
  Asian-East Asian Heritage | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Withdrawal From Study
Description: The time from randomization to the time at which the participant was withdrawn from the Double-Blind Phase of the study for any reason was measured. No data are reported for the Lamotrigine group because of an incalculable confidence interval. See the outcome measure entitled "Number of Participants with a Withdrawal Event" for data regarding the number of participants who withdrew from the study.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: Full Analysis Set in Randomized (double-blind) Phase (FAS2): participants who received at least one dose of study medication in the Randomized Phase (RP) and had at least one post-treatment efficacy assessment in the RP. The upper limit of the confidence interval was not calculable for the Lamotrigine group due to an insufficient number of events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 0
days | 67.5 [32.0 to 127.0] |
Statistical Analysis 1: Comparison: Placebo vs Lamotrigine 200 mg; Test type: Superiority or Other; p = 0.010, Log Rank

2. Secondary Outcome: Time to Intervention for Any Mood Episode (TIME)
Description: The TIME was defined as the time from entry into the Randomized Phase to the time of the first prescription of any additional pharmacotherapy or electroconvulsive therapy (ECT) determined by the Investigator to be necessary for treatment of a relapse or recurrence of depression or the recurrence of a manic, hypomanic, or mixed episode, whichever occurred first. Categorization as a manic, hypomanic, or mixed episode was left to the Investigator's discretion. See the outcome measure entitled "Number of Participants with Intervention for Any Mood Episode" for data related to TIME.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2. In the Lamotrigine 200 mg group, the estimated median TIME was not calculable because the probability of not reaching TIME remained greater than 0.50 throughout the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 0
days | 109.0 [43.0 to 141.0] |

3. Secondary Outcome: Time to Intervention for Depressive Episode (TIDep)
Description: The TIDep was defined as the time from entry into the Randomized Phase to the time of the first prescription of any additional pharmacotherapy or ECT determined by the Investigator to be necessary for treatment of a relapse or recurrence of depression episode. No data are being presented for either treatment group. See the outcome measure entitled "Number of Participants with Intervention for Depressive Episode" for data related to TIDep.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2. In the Lamotrigine 200 mg group, the estimated median TIDep was not calculable because the probability of not reaching TIDep remained greater than 0.50 throughout the study. The upper limit of the confidence interval was not calculable for the Placebo group due to an insufficient number of events.
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Intervention for Manic, Hypomanic, or Mixed Episode (TIMan)
Description: The TIMan was defined as the time from entry into the Randomized Phase to the time of the first prescription of any additional pharmacotherapy or ECT determined by the Investigator to be necessary for treatment of the relapse or recurrence of a manic, hypomanic, or mixed episode. No data are being presented for either treatment group. See the outcome measure entitled "Number of Participants with Intervention for a Manic, Hypomanic, or Mixed Episode" for data related to TIMan.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2. In both groups, the estimated median TIMan was not calculable because the probability of not reaching TIMan remained greater than 0.50 throughout the study.
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinical Global Impressions of Improvement (CGI-I) at Week 26/Withdrawal (Randomized Phase)
Description: The CGI-I is a 7-point scale that assessed the participant's global improvement compared to his/her condition at study entry whether or not, in the judgement of the Investigator, it was due entirely to drug treatment; 0=not assessed, 1= very much improved to 7= very much worse.
Time Frame: Week 26/Withdrawal
Population: FAS2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
points on a scale | 3.5 (1.50) | 2.4 (1.29)

6. Secondary Outcome: Clinical Global Impressions of Improvement (CGI-I) at Week 16/Withdrawal (Preliminary Phase)
Description: as for outcome 5
Time Frame: Week 16/Withdrawal
Population: Full Analysis Set in the Preliminary Phase (FAS1): all participants who received at least one dose of study medication for the Preliminary Phase and underwent at least one efficacy assessment after receiving the study medication in the Preliminary Phase. Nine participants in the Lamotrigine 25-200 mg group have no data for the CGI-I.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Lamotrigine 25-200 mg
Number analyzed (Participants) | 206
points on a scale | 3.1 (1.56)

7. Secondary Outcome: Change From Baseline in Clinical Global Impressions of Severity (CGI-S) Scores at Week 26/Withdrawal (Randomized Phase)
Description: The CGI-S is a 7-point scale that assessed the participant's severity of illness based on the total clinical experience of the Investigator with this particular population; 0=not assessed, 1= normal, not at all ill to 7= among the most extremely ill participants. Change from baseline was calculated as the Week 26/Withdrawal value minus the baseline value (at the time of randomization).
Time Frame: Baseline and Week 26/Withdrawal
Population: FAS2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
points on a scale | 1.0 (1.19) | 0.4 (1.25)

8. Secondary Outcome: Change From Baseline in Clinical Global Impressions of Severity (CGI-S) Scores at Week 16/Withdrawal (Preliminary Phase)
Description: The CGI-S is a 7-point scale that assessed the participant's severity of illness based on the total clinical experience of the Investigator with this particular population; 0=not assessed, 1= normal, not at all ill to 7= among the most extremely ill participants. Change from baseline was calculated as the Week 16/Withdrawal value minus the baseline value (at Week 0 of the Preliminary Phase).
Time Frame: Baseline and Week 16/Withdrawal
Population: FAS1. Nine participants in the Lamotrigine 25-200 mg group have no data for the CGI-S at Week 16/Withdrawal.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Lamotrigine 25-200 mg
Number analyzed (Participants) | 206
points on a scale | -0.7 (1.39)

9. Secondary Outcome: Change From Baseline in Hamilton Rating Scale for Depression (HAMD-17) Scores at Week 26/Withdrawal (Randomized Phase)
Description: The HAMD-17 is a 17-item questionnaire that detects change and measures illness severity. Individual items are rated on a scale of 0-4, 0-3, and 0-2 with the total HAMD-17 score ranging from 0 (not ill) to 52 (severely ill). Change from baseline was calculated as the Week 26/Withdrawal value minus the baseline value (at the time of randomization).
Time Frame: Baseline and Week 26/Withdrawal
Population: FAS2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
points on a scale | 5.4 (7.39) | 2.7 (7.77)

10. Secondary Outcome: Change From Baseline in Hamilton Rating Scale for Depression (HAMD-17) Scores at Week 16/Withdrawal (Preliminary Phase)
Description: The HAMD-17 is a 17-item questionnaire that detects change and measures illness severity. Individual items are rated on a scale of 0-4, and 0-2, with the total HAMD-17 score ranging from 0 (not ill) to 52 (severely ill). Change from baseline was calculated as the Week 16/Withdrawal value minus the baseline value (at Week 0 of the Preliminary Phase).
Time Frame: Baseline and Week 16/Withdrawal
Population: FAS1. Nine participants in the Lamotrigine 25-200 mg group have no data for the HAMD-17 at Week 16/Withdrawal.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Lamotrigine 25-200 mg
Number analyzed (Participants) | 206
points on a scale | -4.1 (9.14)

11. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Scores at Week 26/Withdrawal (Randomized Phase)
Description: The YMRS is an 11-item questionnaire that detects change and measures illness severity. Individual items are rated on a scale of 0-8 and 0-4, with the total YMRS score ranging from 0 (not ill) to 60 (severely ill). Change from baseline was calculated as the Week 26/Withdrawal value minus the baseline value (at the time of randomization).
Time Frame: Baseline and Week 26/Withdrawal
Population: FAS2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
points on a scale | 2.2 (6.59) | 1.0 (5.67)

12. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Scores at Week 16/Withdrawal (Preliminary Phase)
Description: The YMRS is an 11-item questionnaire that detects change and measures illness severity. Individual items are rated on a scale of 0-8 and 0-4, with the total YMRS score ranging from 0 (not ill) to 60 (severely ill). Change from baseline was calculated as the Week 16/Withdrawal value minus the baseline value (at Week 0 of the Preliminary Phase).
Time Frame: Baseline and Week 16/Withdrawal
Population: FAS1. Nine participants in the Lamotrigine 25-200 mg group have no data for the HAMD-17 at Week 16/Withdrawal.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Lamotrigine 25-200 mg
Number analyzed (Participants) | 206
points on a scale | 0.4 (10.45)

13. Post Hoc Outcome: Number of Participants With a Withdrawal Event
Description: The number of participants who withdrew from the study was measured. This outcome measure was added post-hoc because no data are being reported for the Lamotrigine group regarding time to study withdrawal. See the primary outcome measure for time to study withdrawal data for the Placebo group. Data from participants who had not withdrawn were defined as censored.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2
Measure: Number; unit: participants
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
participants
  Withdrawal Event | 43 | 24
  Censored | 15 | 21

14. Post Hoc Outcome: Number of Participants With Intervention for Any Mood Episode
Description: The number of participants with intervention for any mood episode was measured. The necessity of the intervention was determined by the Investigator's discretion. This outcome measure was added post-hoc because no data are being reported for the Lamotrigine group regarding time to intervention for any mood episode (TIME). See the outcome measure for TIME for data for the Placebo group. Data from participants who had not met TIME were defined as censored.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2
Measure: Number; unit: participants
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
participants
  Intervention Event | 37 | 20
  Censored | 21 | 25

15. Post Hoc Outcome: Number of Participants With Intervention for Depressive Episode
Description: The number of participants with intervention for depressive episode was measured. The necessity of the intervention was determined by the Investigator's discretion. This outcome measure was added post-hoc because no data are being reported for the Placebo or Lamotrigine groups regarding time to intervention for depressive episode (TIDep). Data from participants who had not met TIDep were defined as censored.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2
Measure: Number; unit: participants
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
participants
  Intervention Event | 27 | 15
  Censored | 31 | 30

16. Post Hoc Outcome: Number of Participants With Intervention for a Manic, Hypomanic, or Mixed Episode
Description: The number of participants with intervention for a manic, hypomanic, or mixed episode was measured. The necessity of the intervention was determined by the Investigator's discretion. This outcome measure was added post-hoc because no data are being reported for the Placebo or Lamotrigine groups regarding time to intervention for manic, hypomanic, or mixed episode (TIMan). Data from participants who had not met TIMan were defined as censored.
Time Frame: Randomization to Study Withdrawal (up to Week 26)
Population: FAS2
Measure: Number; unit: participants
Arm/Group | Placebo | Lamotrigine 200 mg
Number analyzed (Participants) | 58 | 45
participants
  Intervention Event | 10 | 5
  Censored | 48 | 40

ADVERSE EVENTS:
Description: Adverse events (AEs) and serious adverse events (SAEs) were collected in the Safety Population (SP). The SP is defined for the Preliminary and Randomized Phases as all participants who received at least one dose of study medication for each phase.
Arm/Group | Lamotrigine 25-200 mg | Placebo | Lamotrigine 200 mg
Serious Adverse Events (participants affected / at risk) | 14/215 | 1/58 | 1/45
Other Adverse Events (participants affected / at risk) | 84/215 | 17/58 | 15/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine 25-200 mg (N=215) | Placebo (N=58) | Lamotrigine 200 mg (N=45)
Mania (Psychiatric disorders) | 8 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 2 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0
Suicide ideation (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine 25-200 mg (N=215) | Placebo (N=58) | Lamotrigine 200 mg (N=45)
Nasopharyngitis (Infections and infestations) | 49 | 13 | 11
Headache (Nervous system disorders) | 22 | 2 | 2
Nausea (Gastrointestinal disorders) | 17 | 2 | 0
Dizziness (Nervous system disorders) | 16 | 1 | 1
Constipation (Gastrointestinal disorders) | 11 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.